CLINICAL TRIAL: NCT02933580
Title: A Double-blind, Placebo-controlled, Randomized, Phase 1, Single Ascending Dose Study to Investigate Safety, Tolerability, and Pharmacokinetics of JNJ-56136379 in Healthy Japanese Adult Subjects
Brief Title: A Study to Investigate Safety, Tolerability, and Pharmacokinetics of JNJ-56136379 in Healthy Japanese Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108247; 56136379HPB1003 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2016-10-12; First posted 2016-10-14 (Estimated); Last update posted 2018-03-16 (Actual); Status verified 2018-03

CONDITIONS: Healthy
MeSH Terms: interventions — JNJ-56136379

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (4):
- Cohort A: JNJ-56136379 (25 mg) or Placebo (Experimental): Participants will receive a single oral dose of 25 milligram (mg) of JNJ-56136379 (1*25-mg tablet) or placebo on Day 1, fasted conditions.
  Interventions: Drug: JNJ-56136379; Other: Placebo
- Cohort B: JNJ-56136379 (150 mg) or Placebo (Experimental): Participants will receive a single oral dose of 150 mg of JNJ-56136379 (2* 25-mg tablet and 1*100-mg tablet) or placebo on Day 1, fasted conditions.
  Interventions: Drug: JNJ-56136379; Other: Placebo
- Cohort C: JNJ-56136379 (300 mg) or Placebo (Experimental): Participants will receive a single oral dose of 300 mg of JNJ-56136379 (3*100-mg tablet) or placebo on Day 1, fasted conditions.
  Interventions: Drug: JNJ-56136379; Other: Placebo
- Cohort D: JNJ-56136379 (600 mg) or Placebo (Experimental): Participants will receive a single oral dose of 600 mg of JNJ-56136379 (6*100-mg tablet) or placebo on Day 1, fasted conditions.
  Interventions: Drug: JNJ-56136379; Other: Placebo

INTERVENTIONS:
Drug: JNJ-56136379 — Participants will receive a single oral dose (tablets) of JNJ-56136379 on Day 1.
Other: Placebo — Participants will receive matching placebo tablets on Day 1.

SUMMARY:
The purpose of this study is to investigate the safety, tolerability, and pharmacokinetics (PK) of JNJ-56136379 in healthy Japanese adult participants following oral administration of single doses from 25 milligram (mg) up to 600 mg, in fasted conditions.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be a Japanese participant who has resided outside Japan for no more than 10 years and whose parents and grandparents are Japanese as determined by participant's verbal report
* Participant must be healthy on the basis of a medical evaluation that reveals the absence of any clinically relevant abnormality and includes a physical examination, medical and surgical history, vital signs, and the results of blood biochemistry, blood coagulation, and hematology tests and a urinalysis performed at screening. If there are abnormalities, the participant may be included only if the investigator judges the abnormalities to be not clinically significant or to be appropriate and reasonable for the population under study. This determination must be recorded in the participant's source documents and initialed/signed by the investigator
* Participant must have a body mass index (BMI; weight in kilogram [kg] divided by the square of height in meters) of 18.0 to 30.0 kilogram per meter square [kg/m^2], extremes inclusive, and body weight not less than 45.0 kg
* Participant must have a normal 12-lead electrocardiogram (ECG) (based on the mean value of the triplicate parameters) at screening including: normal sinus rhythm (heart rate between 45 and 100 beats per minute [bpm], extremes included); QT interval corrected for heart rate according to Fridericia (QTcF) less than or equal to (<=)450 millisecond (ms); QRS interval less than (<)120 ms; PR interval <=220 ms
* A female participant (except if permanently sterile), should have a negative serum pregnancy test at screening and all female participants should have a negative urine pregnancy test on Day -1

Exclusion Criteria:

* Participant with a past history of cardiac arrhythmias (example [eg], extrasystoli, tachycardia at rest), history of risk factors for Torsade de Pointes syndrome (eg, hypokalemia, family history of long QT Syndrome)
* Female participant who is breastfeeding at screening or pregnant at screening or predose
* Male participant planning to father a child while enrolled in this study or within 90 days after study drug administration
* Participant with current human immunodeficiency virus type 1 (HIV-1) or HIV-2 infection (confirmed by antibodies) at Screening
* Participant with current hepatitis A infection (confirmed by hepatitis A antibody immunoglobulin M [IgM]), or hepatitis B virus (HBV) infection (confirmed by HBsAg), or hepatitis C virus (HCV) infection (confirmed by HCV antibody), or hepatitis E infection (confirmed by hepatitis E antibody IgM) at Screening

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2016-10-12 (Actual); Primary Completion 2017-02-04 (Actual); Study Completion 2017-02-04 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | Up to 29 days
  The Cmax is the maximum observed plasma concentration.
Time to Reach Maximum Observed Plasma Concentration (Tmax) | Up to 29 days
  The Tmax is defined as actual sampling time to reach maximum observed plasma analyte concentration.
Area Under the Concentration-Time Curve from time 0 to the Time of the Last Measurable non-Below Quantification Limit Concentration (AUC [0-last]) | Up to 29 days
  AUC (0-last) is defined as area under the analyte concentration-time curve from time 0 to the time of the last measurable (non-below quantification limit [BQL]) concentration, calculated by linear-linear trapezoidal summation.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC [0-infinity]) | Up to 29 days
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC(last) and C(last)/lambda(z); wherein AUC(last) is area under the plasma concentration-time curve from time zero to last observed measurable (non-BQL) concentration, and lambda(z) is elimination rate constant; extrapolations of more than 20.00 percent (%) of the total AUC are reported as approximations.
Number of Participants With Adverse events as a Measure of Safety and Tolerability | 30-35 days after study drug intake (approximately 8 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Glendale, California, United States